CLINICAL TRIAL: NCT00099359
Title: Phase III Randomized Trial of the Safety and Efficacy of Three Neonatal Antiretroviral Regimens for Prevention of Intrapartum HIV-1 Transmission
Brief Title: Trial of Three Neonatal Antiretroviral Regimens for Prevention of Intrapartum HIV Transmission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NICHD/HPTN 040 (P1043)
Record Dates: First submitted 2004-12-10; First posted 2004-12-13 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2011-02

CONDITIONS: Disease Transmission, Vertical; Vertical Human Immunodeficiency Virus Transmission; HIV Infections
Keywords: HIV; Perinatal; Prevention; Transmission; Nevirapine; Epivir; Zidovudine; Nelfinavir; ZDV; NVP; 3TC; NFV; Viracept; Viramune; HIV Seronegativity; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Nevirapine; Lamivudine; Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Standard of care ( Zidovudine only)
  Interventions: Drug: Zidovudine
- B (Experimental): Standard of care (Zidovudine) plus Nevirapine
  Interventions: Drug: Nevirapine (NVP)
- C (Experimental): Standard of Care (Zidovudine) plus 2 weeks of Epivir and Nelfinavir
  Interventions: Drug: Epivir (3TC); Drug: Nelfinavir (NFV)

INTERVENTIONS:
Drug: Zidovudine — Given for 6 weeks. 12mg PO BID if birthweight (BW) > 2000 grams 8 mg PO BID if BW < 2000 grams
  Other Names: Retrovir
  Arms: A
Drug: Nevirapine (NVP) — Standard of Care (Zidovudine) plus
  NVP, first dose initiated within 48 hrs of birth, second dose 48 hrs (+ 4 hours) after the first dose, and third dose 96 hours (+ 4 hours) after the second dose :
  12 mg PO per dose if BW > 2000 grams, 8 mg PO per dose if BW < 2000 grams
  Other Names: Viramune
  Arms: B
Drug: Epivir (3TC) — Stand of care (Zidovudine) plus
  3TC, given for 2 weeks: 6 mg po bid if BW > 2000 grams 4 mg po bid if BW < 2000 grams AND
  NFV, given for 2 weeks:
  200 mg po bid if BW > 3000 grams 150 mg po bid if BW > 2,000 - 3000 grams 100 mg PO BID if BW < 2000 grams
  Other Names: Lamivudine
  Arms: C
Drug: Nelfinavir (NFV) — 200 mg BID if birth weight (BW) > 3000 grams for 2 weeks;150 mg BID if BW > 2000-3000 grams for 2 weeks; 100 mg BID BW </= 2000 grams for 2 weeks
  Other Names: Viracept
  Arms: C

SUMMARY:
Giving anti-HIV medications to babies born of HIV positive mothers right after birth can lower the babies' risk of contracting HIV. This study will assess the safety and efficacy of two different combinations of anti-HIV medications compared to a one drug standard regimen in preventing mother to baby transmission. The one drug standard treatment and two combinations to be studied are: 1) zidovudine, 2) zidovudine/nevirapine and 3) zidovudine/lamivudine/nelfinavir.

DETAILED DESCRIPTION:
Despite the notable reductions in perinatal transmission of HIV-1 with antiretroviral therapy and other interventions, perinatal transmission continues to occur at rates of 20-30% among pregnant women who are not identified as HIV-1-infected and/or are not provided with antiretroviral therapy. The optimum treatment strategy for prevention of transmission of HIV-1 to infants born to these women is unknown. No trials have evaluated the efficacy of neonatal antiretroviral therapy alone but observational data suggest benefit from zidovudine (ZDV) therapy given to the infant beginning within 48 hours of birth and continued for six weeks. This protocol will compare the safety and efficacy of three antiretroviral regimens administered in the neonatal period: Arm A- ZDV, Arm B- ZDV plus nevirapine (NVP), and Arm C- ZDV plus nelfinavir (NFV) and lamivudine (3TC). Two regimens were selected based on expected antiretroviral activity, pharmacokinetic data, and toxicity profiles. Standard of care (6 weeks of ZDV) alone will be compared to the 6 weeks of ZDV plus either 3 doses of NVP or 2 weeks of 3TC and NFV. Arm B (ZDV + NVP) is the regimen expected to provide the best profile when factors of efficacy, safety, cost, acceptability and convenience are considered. The comparison of Arms B and C is also of considerable interest since the 2-drug Arm B is easier to implement and less expensive than the triple drug Arm C. Although triple drug therapies have been recommended for post-exposure prophylaxis for needle-stick injuries in high-risk circumstances, it is unknown whether the triple drug arm will provide better efficacy than the 2-drug arm for post-exposure prophylaxis of the infant.

This open-label study is expected to accrue 1731 infants of women identified in labor as being HIV positive or who are HIV positive but have not received antiretroviral medication during the pregnancy. If eligible the infant will be randomized at birth to one of three aforementioned treatment arms. Medical history, social, demographic, physical exam, RNA and T- lymphocyte data are collected on the mother during the delivery visit. The infant will have a birth visit and then return for 1-week, 2-week, 4-week, 3-month and a final 6-month visit. Infant evaluations will include: a medical history and physical exam, DNA testing, CBC and liver function tests, cells for long-term storage and RNA/CD4/CD8 testing if HIV positive. The initial study drug doses will be given to the infant while in the hospital. Mothers will administer the infants' remaining treatment doses at home depending on ability.

ELIGIBILITY:
Inclusion Criteria:

Infants who meet all of the following criteria are eligible for the study:

* Mother known to be HIV-1-infected prior to labor or identified at the time of labor or <48 hours postpartum. HIV-1 infection for the purposes of enrollment into this study is defined as: (a) Single positive HIV-1 rapid test in mother or her infant; or (b) Historical documentation of a positive HIV-1 diagnostic test confirmed by repeat diagnostic testing for HIV-1 according to country guidelines in mother (written documentation of test results must be present in the medical record).
* Maternal written informed consent for study participation.
* Mother has not received any antiretroviral therapy during the current pregnancy prior to the onset of labor and delivery; women may have received intravenous or oral ZDV during labor. Women may have received any antiretroviral therapy in previous pregnancies for prevention of vertical HIV-1 transmission.
* Infant is <48 hours old. Infant may have received up to 48 hours of ZDV as standard care before study enrollment.

Exclusion Criteria:

Infants who meet any of the following criteria will be excluded from the study:

* Extreme prematurity (< 32 weeks of gestation).
* Birth weight <1500 grams.
* Presence of life-threatening conditions.
* Inability to take oral medication throughout the first 48 hours of life (must be able to receive oral medication by age 48 hours).
* Maternal inability to provide informed consent because of a lack of a conscious state, psychiatric conditions, or language barriers.
* Mother received any antiretroviral therapy during labor and delivery other than intravenous or oral ZDV.

Max Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1735 (Actual)
Dates: Start 2004-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Nielsen, MD, Study Chair — University of California, Los Angeles
Locations (17):
- United States (5):
  - Miller Children's Hospital, Long Beach, California
  - University of FL, Gainesville, Florida
  - University of FL-HSC, Jacksonville, Florida
  - University Medical and Dental School of NJ-Newark Campus, Newark, New Jersey
  - Texas Childrens Hospital, Houston, Texas
- Hospital I. G. A. Dr. Diego Paroissien, Buenos Aires, Argentina
- Brazil (8):
  - Federal University of Minas Gerais (UFMG), Belo Horizonte, Minas Gerais
  - Universidade de Sao Paulo (USP) , MD, São Paulo, Ribeirão Preto
  - Hospital Fêmina S.A. Unidade Perinatal de Transmissão Vertical, Porto Alegre, Rio Grande do Sul
  - Hospital Santa Casa (HSC), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao (GHC), Porto Alegre, Rio Grande do Sul
  - Hospital dos Servidores do Estado (HSE), Rio de Janeiro
  - Hospital Geral de Novo Iguacu, Rio de Janeiro
  - 5088 - Universidade Federal de Sao Paulo (UFSP), São Paulo
- San Juan Hospital, San Juan, Puerto Rico
- South Africa (2):
  - Tygerberg Hospital, Cape Town
  - Chris Hani Baragwanath Hospital, Johannesburg

REFERENCES:
- [Result] Mirochnick M, Nielsen-Saines K, Pilotto JH, Pinto J, Veloso VG, Rossi S, Moye J, Bryson Y, Mofenson L, Camarca M, Watts DH; NICHD HPTN 040/PACTG 1043 PROTOCOL Team. Nelfinavir and Lamivudine pharmacokinetics during the first two weeks of life. Pediatr Infect Dis J. 2011 Sep;30(9):769-72. doi: 10.1097/INF.0b013e3182242950. PMID 21666540
- [Result] Mirochnick M, Nielsen-Saines K, Pilotto JH, Pinto J, Jimenez E, Veloso VG, Parsons T, Watts DH, Moye J, Mofenson LM, Camarca M, Bryson Y; NICHD/HPTN 040/PACTG 1043 Protocol Team. Nevirapine concentrations in newborns receiving an extended prophylactic regimen. J Acquir Immune Defic Syndr. 2008 Mar 1;47(3):334-7. PMID 18398973
- [Result] Nielsen-Saines K, Watts DH, Veloso VG, Bryson YJ, Joao EC, Pilotto JH, Gray G, Theron G, Santos B, Fonseca R, Kreitchmann R, Pinto J, Mussi-Pinhata MM, Ceriotto M, Machado D, Bethel J, Morgado MG, Dickover R, Camarca M, Mirochnick M, Siberry G, Grinsztejn B, Moreira RI, Bastos FI, Xu J, Moye J, Mofenson LM; NICHD HPTN 040/PACTG 1043 Protocol Team. Three postpartum antiretroviral regimens to prevent intrapartum HIV infection. N Engl J Med. 2012 Jun 21;366(25):2368-79. doi: 10.1056/NEJMoa1108275. PMID 22716975
- [Derived] Adachi K, Xu J, Ank B, Watts DH, Camarca M, Mofenson LM, Pilotto JH, Joao E, Gray G, Theron G, Santos B, Fonseca R, Kreitchmann R, Pinto J, Mussi-Pinhata MM, Machado DM, Ceriotto M, Morgado MG, Bryson YJ, Veloso VG, Grinsztejn B, Mirochnick M, Moye J, Nielsen-Saines K; MPH for the NICHD HPTN 040 Study Team. Congenital Cytomegalovirus and HIV Perinatal Transmission. Pediatr Infect Dis J. 2018 Oct;37(10):1016-1021. doi: 10.1097/INF.0000000000001975. PMID 30216294
- [Derived] Yeganeh N, Watts DH, Xu J, Kerin T, Joao EC, Pilotto JH, Theron G, Gray G, Santos B, Fonseca R, Kreitchmann R, Pinto J, Mussi-Pinhata MM, Veloso V, Camarca M, Mofenson L, Moye J, Nielsen-Saines K. Infectious Morbidity, Mortality and Nutrition in HIV-exposed, Uninfected, Formula-fed Infants: Results From the HPTN 040/PACTG 1043 Trial. Pediatr Infect Dis J. 2018 Dec;37(12):1271-1278. doi: 10.1097/INF.0000000000002082. PMID 29750766
- [Derived] Adachi K, Xu J, Yeganeh N, Camarca M, Morgado MG, Watts DH, Mofenson LM, Veloso VG, Pilotto JH, Joao E, Gray G, Theron G, Santos B, Fonseca R, Kreitchmann R, Pinto J, Mussi-Pinhata MM, Ceriotto M, Machado DM, Bryson YJ, Grinsztejn B, Moye J, Klausner JD, Bristow CC, Dickover R, Mirochnick M, Nielsen-Saines K; NICHD HPTN 040 Study Team. Combined evaluation of sexually transmitted infections in HIV-infected pregnant women and infant HIV transmission. PLoS One. 2018 Jan 5;13(1):e0189851. doi: 10.1371/journal.pone.0189851. eCollection 2018. PMID 29304083
- [Derived] Adachi K, Xu J, Ank B, Watts DH, Mofenson LM, Pilotto JH, Joao E, Santos B, Fonseca R, Kreitchmann R, Pinto J, Mussi-Pinhata MM, Gray G, Theron G, Morgado MG, Bryson YJ, Veloso VG, Klausner JD, Moye J, Nielsen-Saines K; NICHD HPTN 040 Study Team. Cytomegalovirus Urinary Shedding in HIV-infected Pregnant Women and Congenital Cytomegalovirus Infection. Clin Infect Dis. 2017 Aug 1;65(3):405-413. doi: 10.1093/cid/cix222. PMID 28369278
- [Derived] Adachi K, Klausner JD, Bristow CC, Xu J, Ank B, Morgado MG, Watts DH, Weir F, Persing D, Mofenson LM, Veloso VG, Pilotto JH, Joao E, Nielsen-Saines K; NICHD HPTN 040 Study Team. Chlamydia and Gonorrhea in HIV-Infected Pregnant Women and Infant HIV Transmission. Sex Transm Dis. 2015 Oct;42(10):554-65. doi: 10.1097/OLQ.0000000000000340. PMID 26372927
- [Derived] Yeganeh N, Watts HD, Camarca M, Soares G, Joao E, Pilotto JH, Gray G, Theron G, Santos B, Fonseca R, Kreitchmann R, Pinto J, Mussi-Pinhata M, Ceriotto M, Machado DM, Grinzstejn B, Veloso VG, Morgado MG, Bryson Y, Mofenson LM, Nielsen-Saines K; NICHD HPTN 040P1043 Study Team. Syphilis in HIV-infected mothers and infants: results from the NICHD/HPTN 040 study. Pediatr Infect Dis J. 2015 Mar;34(3):e52-7. doi: 10.1097/INF.0000000000000578. PMID 25742089
- See also: home page of the National Institute of Child Health and Human Development — http://www.nichd.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 02/27/2004 and the study ended 02/28/2011. A total of 17 sites in Brazil, South Africa, Argentina and the U.S. participated in the study.
Groups:
- Arm A (ZDV Only): Standard of care ( Zidovudine only). 12 mg PO BID if BW>2000 grams ; 8 mg PO BID if BW</= 2000 grams
- ARM B (ZDV + NVP): Standard of care (Zidovudine) plus Nevirapine (NVP)
  NVP, first dose initiated within 48 hrs of birth, second dose 48 hrs (+ 4 hours) after the first dose, and third dose 96 hours (+ 4 hours) after the second dose :
  12 mg PO per dose if BW > 2000 grams, 8 mg PO per dose if BW < 2000 grams
- ARM C (ZDV + 3TC + NFV): Standard of Care (Zidovudine) plus 2 weeks of Epivir (3TC) and Nelfinavir (NFV) 3TC, given for 2 weeks: 6 mg po bid if BW > 2000 grams 4 mg po bid if BW < 2000 grams AND
  NFV, given for 2 weeks:
  200 mg po bid if BW > 3000 grams 150 mg po bid if BW > 2,000 - 3000 grams 100 mg PO BID if BW < 2000 grams
Period: Overall Study
Arm/Group | Arm A (ZDV Only) | ARM B (ZDV + NVP) | ARM C (ZDV + 3TC + NFV)
Started | 581 | 580 | 574
Completed | 527 | 515 | 506
Not Completed | 54 | 65 | 68
Not completed — Death | 11 | 15 | 17
Not completed — Withdrawal by Subject | 19 | 19 | 23
Not completed — Lost to Follow-up | 15 | 24 | 24
Not completed — moved out of area | 9 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (ZDV Only) | ARM B (ZDV + NVP) | ARM C (ZDV + 3TC + NFV) | Total
Number analyzed (Participants) | 581 | 580 | 574 | 1735
Age Continuous [Mean (Standard Deviation); unit: weeks]
  Gestational Age in Weeks | 39 (1.7) | 39 (1.5) | 39 (1.7) | 39 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 303 | 281 | 882
  Male | 283 | 277 | 293 | 853
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 12
  Puerto Rico | 0 | 1 | 1 | 2
  Argentina | 10 | 6 | 11 | 27
  Brazil | 409 | 408 | 402 | 1219
  South Africa | 158 | 161 | 156 | 475

OUTCOME MEASURES:

1. Primary Outcome: Infant HIV Infection Status
Description: Intrapartum HIV infection at 3 Months
Time Frame: 3 months
Population: All infants with HIV-1 test results except infants infected at birth (i.e. in utero infections) were included in these analysis.
Measure: Number; unit: participants
Groups:
- ARM A (ZDV - Standard of Care): ZDV (standard of care), given for 6 weeks:
  12 mg PO BID if birthweight (BW) > 2000 grams 8 mg PO BID if BW < 2000 grams
- ARM B (ZDV + NVP): plus NVP, first dose initiated within 48 hrs of birth, second dose 48 hrs (+ 4 hours) after the first dose, and third dose 96 hours (+ 4 hours) after the second dose : 12 mg PO per dose if BW > 2000 grams, 8 mg PO per dose if BW < 2000 grams
- ARM C (ZDV +3TC+NFV): ZDV (standard of care) plus 3TC, given for 2 weeks:
  6 mg po bid if BW > 2000 grams 4 mg po bid if BW < 2000 grams AND
  NFV, given for 2 weeks:
  200 mg po bid if BW > 3000 grams 150 mg po bid if BW > 2,000 - 3000 grams 100 mg PO BID if BW < 2000 grams
Arm/Group | ARM A (ZDV - Standard of Care) | ARM B (ZDV + NVP) | ARM C (ZDV +3TC+NFV)
Number analyzed (Participants) | 566 | 562 | 556
participants | 24 | 11 | 12
Statistical Analysis 1: Comparison: ARM A (ZDV - Standard of Care) vs ARM B (ZDV + NVP) vs ARM C (ZDV +3TC+NFV); Test type: Superiority or Other; p = .046, multiple comparison — Overall comparison of 3 KM curves using an extension of the M-H test was performed. Results indicated a significant difference therefore a 2nd stage analysis was done to compare each pair of transmission rates, using 2-sample Mantel-Haenzel tests; Hochberg's modified Bonferroni method was used to adjust the significance level for comparisons between arms

2. Primary Outcome: Participants With Serious Adverse Events
Description: Serious Adverse Events by System Organ Class=Blood and lymphatic system disorders
Time Frame: through age 6 months.
Measure: Number; unit: participants
Groups:
- ARM A (ZDV Only): ZDV only
- ARM B (ZDV + NVP): ZDV + NVP
- ARM C (ZDV + 3TC/NFV): ZDV + 3TC/NFV
Arm/Group | ARM A (ZDV Only) | ARM B (ZDV + NVP) | ARM C (ZDV + 3TC/NFV)
Number analyzed (Participants) | 566 | 562 | 556
participants | 86 | 59 | 110
Statistical Analysis 1: Comparison: ARM A (ZDV Only) vs ARM B (ZDV + NVP) vs ARM C (ZDV + 3TC/NFV); Test type: Superiority or Other; p = .0001, Chi-squared

3. Secondary Outcome: Infant HIV-1 Infection Status
Description: In utero HIV-1 infection rate
Time Frame: birth
Measure: Number; unit: participants
Arm/Group | Arm A (ZDV Only) | ARM B (ZDV + NVP) | ARM C (ZDV + 3TC + NFV)
Number analyzed (Participants) | 581 | 580 | 574
participants | 37 | 28 | 28
Statistical Analysis 1: Comparison: Arm A (ZDV Only) vs ARM B (ZDV + NVP) vs ARM C (ZDV + 3TC + NFV); Test type: Superiority or Other; p = .2432, multiple comparison

4. Secondary Outcome: Participant Deaths
Time Frame: through age 6 months
Measure: Number; unit: participants
Arm/Group | Arm A (ZDV Only) | ARM B (ZDV + NVP) | ARM C (ZDV + 3TC + NFV)
Number analyzed (Participants) | 581 | 580 | 574
participants | 11 | 15 | 17
Statistical Analysis 1: Comparison: Arm A (ZDV Only) vs ARM B (ZDV + NVP) vs ARM C (ZDV + 3TC + NFV); Test type: Superiority or Other; p = 0.49, Chi-squared

5. Secondary Outcome: Clinical Covariates of HIV-1 Infection
Description: Compare HIV-1 RNA levels; CD4+ lymphocyte counts; and rates of genotypic and phenotypic resistance among the three treatment regimens.
Time Frame: through age 3 months
Reporting Status: Not Posted

6. Secondary Outcome: 3TC and NFV Pharmacokinetics
Description: Descriptive study of 3TC and NFV pharmacokinetics during first two weeks of life using weight band dosing regimen in a subset of enrolled infants.
Time Frame: through age 14 days
Population: This was a descriptive study. A total of 26 infants were analyzed with 14 at age 4-7 days and 12 at 10-14 days.Plasma samples were collected prior to first AM dose and then at 1,2,4,8 and 12 hours.
Measure: Median (Full Range); unit: ug*h/mL
Groups:
- ARM C (ZDV + 3TC/NFV): Standard ZDV for 6 weeks combined with 2 weeks of 3TC and NFV. NFV and 3TC plasma concentrations were measured by validated HPLC assays with lower detection limit of 0.04 micrograms/mL.
Arm/Group | ARM C (ZDV + 3TC/NFV)
Number analyzed (Participants) | 26
ug*h/mL
  (NFV-AUC-12h) 4-7 day | 20.7 (46.57) [3.4 to 183.5]
  (NFV-AUC-12h) 10-14 day | 25.5 (13.10) [1.7 to 41.7]
  (3TC-AUC-12 h) 4-7 day | 4.0 (4.50) [2.9 to 15.6]
  (3TC-AUC-12h) 10-14 day | 7.9 (4.12) [2.7 to 14]

7. Secondary Outcome: Risk Factors for Perinatal HIV-1 Transmission
Description: Risk factors to be assessed include maternal HIV-1 RNA levels at delivery, maternal syphilis and other infections, obstetrical factors such as duration of membrane rupture, and adherence to neonatal medication.
Time Frame: through age 3 months
Population: All available demographic and clinical variables were tested for association with transmission rate. All variables that were significant at p ≤ 0.20 were included in the multivariable regression model. Variables that were not significant were then removed from the model. The backward elimination method was used to select the final model.
Measure: Number; unit: participants
Groups:
- Infected: Infants infected after birth
- Uninfected: Infants uninfected after birth
Arm/Group | Infected | Uninfected
Number analyzed (Participants) | 47 | 1544
participants
  Treatment Arm C (ZDV+3TC/NFV) | 12 | 516
  Treatment Arm B (ZDV+NFV) | 11 | 523
  Treatment Arm A (ZDV only) | 24 | 505
  Illegal Substance Abuse during pregnancy | 7 | 130
Statistical Analysis 1: Comparison: Infected vs Uninfected; Test type: Superiority or Other; p = 0.05, Regression, Logistic; Adjusted Odds ratio for treatment arm C (ZDV+3TC/NFV) association with Intrapartum Infection Status with Treatment Arm A (ZDV only) as reference group; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.24 to 1.01]
Statistical Analysis 2: Comparison: Infected vs Uninfected; Test type: Superiority or Other; p = 0.01, Regression, Logistic — Adjusted odds ratio for association of treatment arm B (ZDV+NVP) with intrapartum infection status with Treatment Arm A (ZDV only) as reference; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.19 to 0.82]
Statistical Analysis 3: Comparison: Infected vs Uninfected; Test type: Superiority or Other; p = 0.03, Regression, Logistic; Adjusted odds ratio for association of illegal substance use during pregnancy and intrapartum HIV infection status with "NO" being reference group; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.08 to 5.86]
Statistical Analysis 4: Comparison: Infected vs Uninfected; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Adjusted odds ratio for the association of continuous log10 viral load with intrapartum infection status; Odds Ratio (OR) = 2.28, 95% CI 2-sided [1.56 to 3.35]

8. Secondary Outcome: NVP Pharmacokinetics
Description: Descriptive study of NVP pharmacokinetics during first two weeks of life using weight band dosing in a subset of enrolled infants.
Time Frame: 14 days
Measure: Median (Full Range); unit: ng/mL
Groups:
- ARM B (ZDV + NVP): NVP concentrations were measured in 14 infants immediately before the 3rd dose, 4 hours post dose, 1 day post dose, 3-5 days post dose and 7 days post dose.
Arm/Group | ARM B (ZDV + NVP)
Number analyzed (Participants) | 14
ng/mL
  NVP conc prior to 3rd dose | 362 [165 to 1728]
  NVP peak conc (Cmax) post 3rd dose | 2286 [1241 to 3811]
  NVP conc 3-5 day post 3rd dose | 459 [73 to 1747]
  NVP conc 7 day post 3rd dose | 76 [25 to 652]

ADVERSE EVENTS:
Time Frame: through 6 months
Description: AE data collected from study entry to off study period
Groups:
- ARM A (ZDV Alone): ZDV, given for 6 weeks:
  12 mg PO BID if birthweight (BW) > 2000 grams 8 mg PO BID if BW < 2000 grams
- ARM B (ZDV + NVP): ZDV, given for 6 weeks:
  12 mg PO BID if birthweight (BW) > 2000 grams 8 mg PO BID if BW < 2000 grams
  AND NVP, first dose initiated within 48 hrs of birth, second dose 48 hrs (+ 4 hours) after the first dose, and third dose 96 hours (+ 4 hours) after the second dose :
  12 mg PO per dose if BW > 2000 grams, 8 mg PO per dose if BW < 2000 grams
- ARM C (ZDV + 3TC/NFV): ZDV, given for 6 weeks:
  12 mg PO BID if birthweight (BW) > 2000 grams 8 mg PO BID if BW < 2000 grams AND 3TC, given for 2 weeks: 6 mg po bid if BW > 2000 grams 4 mg po bid if BW < 2000 grams AND
  NFV, given for 2 weeks:
  200 mg po bid if BW > 3000 grams 150 mg po bid if BW > 2,000 - 3000 grams 100 mg PO BID if BW < 2000 grams
Arm/Group | ARM A (ZDV Alone) | ARM B (ZDV + NVP) | ARM C (ZDV + 3TC/NFV)
Serious Adverse Events (participants affected / at risk) | 219/581 | 211/580 | 252/574
Other Adverse Events (participants affected / at risk) | 492/581 | 482/580 | 480/574
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A (ZDV Alone) (N=581) | ARM B (ZDV + NVP) (N=580) | ARM C (ZDV + 3TC/NFV) (N=574)
Anaemia Nos (Blood and lymphatic system disorders) | 48 (51) | 28 (32) | 39 (46)
Axillary Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Isoimmune Haemolytic Disease (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 33 (34) | 33 (40) | 71 (83)
Polycythaemia Nos (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocythaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 9 (10)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cyanosis Nos (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Valve Stenosis (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Tachycardia Nos (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tricuspid Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Disorder Nos (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Nos (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Congenital Atrial Septal Defect (Congenital, familial and genetic disorders) | 5 (5) | 4 (4) | 4 (4)
Congenital Cardiac Septal Defect Nos (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Congenital Choroid Plexus Cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Congenital Clubfoot (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1)
Congenital Cytomegalovirus Infection (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Congenital Infection Nos (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Congenital Macrocephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Congenital Syphilis (Congenital, familial and genetic disorders) | 47 (47) | 52 (52) | 42 (43)
Congenital Toxoplasmosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Congenital Ventricular Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 2 (2)
Foetal Alcohol Syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Genitalia External Ambiguous (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Meningomyelocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) | 1 (1)
Retinoblastoma Nos (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 1 (1)
Urethral Valves (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Neonatal Conjunctivitis Nos (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Acquired Pyloric Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea Nos (Gastrointestinal disorders) | 4 (4) | 4 (4) | 6 (6)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Obstruction Nos (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Perforation Nos (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting Nos (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Drug Withdrawal Syndrome Neonatal (General disorders) | 1 (1) | 1 (1) | 0 (0)
Multi-Organ Failure (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 5 (5) | 1 (1)
Sudden Infant Death Syndrome (General disorders) | 1 (1) | 2 (2) | 5 (5)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1)
Jaundice Nos (Hepatobiliary disorders) | 10 (10) | 3 (3) | 2 (2)
Abscess Nos (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Breast Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 13 (14) | 28 (30) | 15 (17)
Bronchitis Acute Nos (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia Nos (Infections and infestations) | 3 (3) | 9 (9) | 8 (9)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis Gangrenous (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis Infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Febrile Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Nos (Infections and infestations) | 21 (24) | 19 (21) | 16 (18)
Gastrointestinal Infection Nos (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Impetigo Nos (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Lobar Pneumonia Nos (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection Nos (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Meningitis Pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neonatal Infection Nos (Infections and infestations) | 5 (5) | 1 (1) | 2 (2)
Omphalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Otitis Media Acute Nos (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Parainfluenzae Virus Infection Nos (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis Carinii Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis Carinii Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Pneumonia Nos (Infections and infestations) | 22 (23) | 17 (17) | 18 (19)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Respiratory Syncytial Virus Infection Nos (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection Nos (Infections and infestations) | 2 (2) | 4 (4) | 2 (2)
Scabies Infestation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis Neonatal (Infections and infestations) | 5 (5) | 3 (3) | 4 (4)
Sepsis Nos (Infections and infestations) | 21 (21) | 16 (18) | 23 (24)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis Nos (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Umbilical Cord Sepsis Nos (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection Nos (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Urinary Tract Infection Nos (Infections and infestations) | 0 (0) | 4 (4) | 3 (3)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Acoustic Stimulation Tests Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 12 (13) | 7 (8) | 5 (6)
Aspartate Aminotransferase Increased (Investigations) | 14 (15) | 7 (8) | 11 (13)
Blood Calcium Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Potassium Increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood Urea Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac Murmur Nos (Investigations) | 0 (0) | 0 (0) | 1 (1)
General Physical Condition Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 2 (2) | 3 (3)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Feeding Problem In Newborn (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
General Nutrition Disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia Nos (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia Nos (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Malnutrition Nos (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Marasmus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic Acidosis Nos (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Underweight (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Tongue Neoplasm Nos (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebral Thrombosis Nos (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsions Nos (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Encephalitis Nos (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Poor Sucking Reflex (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Visual Field Defect Nos (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice Neonatal (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 3 (3) | 6 (6)
Premature Baby (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 6 (6) | 10 (10)
Small For Dates Baby (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 9 (9)
Renal Failure Nos (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma Nos (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis Nos (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchospasm Nos (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cyanosis Neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neonatal Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Obstructive Airways Disorder Nos (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pneumothorax Nos (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Artery Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Oedema Nos (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Face Oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria Nos (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Exposure To Communicable Disease (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Social Problem Nos (Social circumstances) | 12 (12) | 14 (14) | 24 (24)
Cardiac Operation Nos (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Eye Excision (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypertension Nos (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasculitis Nos (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A (ZDV Alone) (N=581) | ARM B (ZDV + NVP) (N=580) | ARM C (ZDV + 3TC/NFV) (N=574)
Anaemia NOS (Blood and lymphatic system disorders) | 286 (451) | 270 (402) | 287 (456)
neutropenia (Blood and lymphatic system disorders) | 225 (294) | 119 (261) | 244 (334)
oral candidiasis (Infections and infestations) | 162 (188) | 170 (194) | 156 (177)
Aspartate Aminotransferase Increased (Investigations) | 335 (439) | 317 (429) | 325 (418)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No